CLINICAL TRIAL: NCT01233479
Title: Immunologic Profile of Patients With Newly Diagnosed Medulloblastoma at Initial Diagnosis and During Standard Radiation and Chemotherapy
Brief Title: Biomarkers in Blood Samples From Young Patients With Newly Diagnosed Brain Tumors Undergoing Standard Radiation Therapy and Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This non-therapeutic study was registered in error. The PRS team doesn't delete studies once registered, so they recommended changing the status to Withdrawn
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett, Pediatric Brain Tumor Consortium
Masking: None | Purpose: Basic Science
Other Study IDs: CDR0000673892; PBTC-N11
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma; untreated childhood cerebellar astrocytoma; untreated childhood cerebral astrocytoma; untreated childhood brain stem glioma; childhood medulloepithelioma; childhood infratentorial ependymoma; newly diagnosed childhood ependymoma; childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Rhabdoid Tumor | interventions — Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: systemic chemotherapy
Other: laboratory biomarker analysis
Procedure: therapeutic surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving radiation therapy and chemotherapy may help doctors learn more about the effects of this treatment on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying biomarkers in blood samples from young patients with newly diagnosed brain tumors undergoing standard radiation therapy and chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the fraction of peripherally circulating T-regulatory cells (T_regs) in pediatric patients with newly diagnosed medulloblastoma and compare it to the levels found in a control group of patients undergoing craniectomy for Chiari malformation.
* Evaluate the longitudinal effects of standard radiotherapy and chemotherapy regimens on the overall population of lymphocytes as well as the fraction of T_reg cells in patients with medulloblastoma.

Secondary

* Determine the baseline fraction of T_reg cells in those with non-medulloblastoma posterior fossa tumors compared to levels found in patients undergoing decompression for Chiari malformation.

OUTLINE: This is a multicenter study.

Patients with Chiari malformation and patients with posterior fossa tumor undergo standard surgery. Patients with posterior fossa tumor also receive standard radiotherapy and chemotherapy.

Blood samples are collected at baseline and periodically to measure the level of circulating T-regulatory cells.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically confirmed posterior fossa tumor

    * Newly diagnosed disease
    * Medulloblastoma OR non-medulloblastoma (pilocytic astrocytoma, ependymoma, atypical rhabdoid tumor, or others)
    * Scheduled to undergo craniotomy and tumor resection
  * Chiari malformation

    * Requires craniectomy for decompression

      * No secondary decompression

PATIENT CHARACTERISTICS:

* No unexplained febrile illness
* No active infection
* No autoimmune disorders such as inflammatory bowel disease, juvenile rheumatoid arthritis, or systemic lupus erythematosus
* No other immunosuppressive disorders (e.g., HIV infection)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Estimated); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Peripherally circulating T-regulatory (T-reg) cells in patients with medulloblastoma or Chiari malformation
Longitudinal side effects of standard radiotherapy and chemotherapy regimens on the overall population of lymphocytes as well as the fraction of circulating T-reg cells
Effect of treatment on lymphocytes and T-reg cells

SECONDARY OUTCOMES:
Baseline fraction of circulating T-reg cells

CONTACTS AND LOCATIONS:
Overall Officials: Sri Gururangan, MD, Principal Investigator — Duke Cancer Institute
Locations (11):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - NCI - Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas